Boiled Peanut Oral Immunotherapy for the Treatment of Peanut Allergic Pediatric Patients

NCT04090203

Study Protocol v3 2/12/2020

# Boiled Peanut Oral Immunotherapy for the Treatment of Peanut Allergic Pediatric Patients (BPOIT)

CCF IRB Number: 18-1294

NCT number: 04090203

IND: 18661

Funded by: Cleveland Clinic RPC
Mark Lauer Pediatric Research Grant

### **Principal Investigator**

Jaclyn Bjelac, MD 9500 Euclid Avenue A120 Cleveland, OH 44195 Bjelacj2@ccf.org 216.445.1449 office 216.316.2754 mobile

### **Co-Investigator/ IND Sponsor**

Alton Melton, MD meltona@ccf.org 216.444.6817

### **Co-Investigator**

Kara McNamara, MD 216.444.4828 mcnamak@ccf.org

### **Co-Investigator**

Leigh Ann Kerns, MD 216.444.6340 Kernsl2@ccf.org

### INVESTIGATOR'S SIGNATURE PAGE

Protocol Amendment: 3

Protocol Date: 12 February 2020

### **Boiled Peanut Oral Immunotherapy for the Treatment of Peanut Allergic Pediatric Patients**(BPOIT)

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable US federal regulations and ICH guidelines.

The trial will be carried out in accordance with International Conference on Harmonization Good Clinical Practice (ICH GCP) and the following:

• United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, and 21 CFR Part 312)

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the Pediatric Research Review Committee (PRRC) and Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. In addition, all changes to the consent form will be IRB-approved; a determination will be made regarding whether a new consent needs to be obtained from participants who provided consent, using a previously approved consent form.

Cleveland, Ohio 44195

Melton/Bjelac 02-12-2020 Amendment #3

### **Table of Contents**

| | Investigator Signature Page & Statement of Compliance | 2 |
|---|---|---|
| 1 | Protocol Summary | 5 |
| 1.1 | Synopsis | 5 |
| 1.2 | Schema | 8 |
| 1.3 | Schedule of Activities | 9 |
| 2 | Introduction | 10 |
| 2.1 | Study Rationale | 10 |
| 2.2 | Background | 10 |
| 2.3 | Risk Benefit Assessment | 13 |
| 3 | Objectives and Endpoints | 15 |
| 4 | Study Design | 17 |
| 4.1 | Overall Design | 17 |
| 4.2 | Scientific Rationale for Study Design | 17 |
| 4.3 | Justification for Dose | 17 |
| 4.4 | End of Study Definition | 17 |
| 5 | Study Population | 18 |
| 5.1 | Inclusion Criteria | 18 |
| 5.2 | Exclusion Criteria | 18 |
| 5.3 | Lifestyle Considerations | 19 |
| 5.4 | Screen Failures | 19 |
| 5.5 | Strategies for Recruitment and Retention | 19 |
| 6 | Study Intervention | 20 |
| 6.1 | Study Intervention Administration | 20 |
| 6.1.1 | Study Intervention Description | 20 |
| 6.1.2 | Dosing and Administration | 22 |
| 6.2 | Preparation/Handling/Storage/Accountability | 27 |
| 6.3 | Measures to Minimize Bias | 28 |
| 6.4 | Study Intervention Compliance | 29 |
| 6.5 | Concomitant Therapy | 29 |
| 6.5.1 | Rescue Medication | 29 |
| 7 | Study Intervention Discontinuation and Participant Discontinuation/Withdrawal | 32 |
| 7.1 | Discontinuation of Study Intervention | 32 |
| 7.2 | Participant Discontinuation/Withdrawal from the Study | 32 |
| 7.3 | Lost to Follow Up | 32 |
| 8 | Study Assessments and Procedures | 34 |
| 8.1 | Efficacy Assessments | 34 |
| 8.2 | Safety and Other Assessments | 34 |
| 8.3 | Adverse Events and Serious Adverse Events | 34 |
| 8.3.1 | Definition of Adverse Events (AEs) | 34 |
| 8.3.2 | Definition of Serious Adverse Events (SAEs) | 34 |
| 8.3.3 | Classification of an Adverse Event | 35 |
| 8.3.4 | Time Period and Frequency for Event Assessment and Follow Up | 35 |
| 8.3.5 | Adverse Event Reporting | 37 |
| 8.3.6 | Serious Adverse Event Reporting | 37 |
| 8.3.7 | Reporting Events to Participants | 37 |

| 8.3.8 | Events of Special Interest | 37 |
|---|---|---|
| 8.3.9 | Reporting of Pregnancy | 38 |
| 8.4 | Unanticipated Problems | 38 |
| 8.4.1 | Definition of Unanticipated Problems | 38 |
| 8.4.2 | Unanticipated Problem Reporting | 38 |
| 8.4.3 | Reporting Unanticipated Problems to Participants | 38 |
| 9 | Statistical Considerations | 39 |
| 9.1 | Statistical Hypotheses | 39 |
| 9.2 | Sample Size Determination | 39 |
| 9.3 | Population for Analyses | 39 |
| 9.4 | Statistical Analysis | 39 |
| 10 | Supporting Documentation and Operational Considerations | 40 |
| 10.1 | Regulatory, Ethical, and Study Oversight Considerations | 40 |
| 10.1.1 | Informed Consent Process | 40 |
| 10.1.1.1 | Consent/Assent and Other Informational Documents Provided to Participants | 40 |
| 10.1.1.2 | Consent Procedures and Documentation | 40 |
| 10.1.2 | Study Discontinuation and Closure | 40 |
| 10.1.3 | Confidentiality and Privacy | 41 |
| 10.1.4 | Future Use of Stored Specimens and Data | 41 |
| 10.1.5 | Key Roles and Governance | 41 |
| 11 | References | 43 |
| 12 | Supplements | 42 |
| 12.1 | Food Allergy Quality of Life Questionnaire for Parents (1-12 years old) | 42 |
| 12.2 | Food Allergy Quality of Life Questionnaire for Parents (13-16 years old) | 43 |
| 12.3 | Dosing/Adverse Event Recording Sheet | 44 |
| 13 | Summary of Changes Table | 45 |

### 1. Protocol Summary

### 1.1 Study Synopsis

**Endpoints:** 

| Title:<br>Study Description: |
|------------------------------|
| Objectives: |

Boiled Peanut Oral Immunotherapy Prospective Phase 1 clinical trial providing proof of concept data on boiled peanut oral immunotherapy (OIT) for the treatment of peanut allergy in children. We hypothesize that the proportion of subjects successfully desensitized with boiled peanut OIT is greater than the theoretical placebo rate of 20%.

- Determine the effect of boiled peanut immunotherapy on the immune response to peanut.
- Compare the safety and tolerability of boiled peanut oral immunotherapy to published data on roasted peanut oral immunotherapy in pediatric subjects with confirmed IgE mediated peanut allergy.
- Primary endpoint: Response to treatment defined as ability to successfully consume a single dose of 300 mg or greater of peanut protein with no dose limiting symptoms at exit double blind placebo controlled food challenge (DBPCFC).
- Secondary endpoints:
- Maximum dose achieved with no or minimal symptoms at exit DBPCFC.
- Change in the maximum tolerated dose from screening to exit DBPCFC.
- The rate of side effects of treatment defined as oral itching, rhinorrhea, conjunctivitis, urticaria, angioedema, abdominal upset, vomiting, diarrhea, cough, wheeze, or anaphylaxis.
- Change in quality of life scores before and after treatment utilizing validated, age specific, food-related quality-of-life surveys before and after peanut oral immunotherapy (Supplement 1)
- Peanut protein component panel, to determine the presence of high levels of sensitivity to peanut proteins known to be associated with severe systemic reactions (Arah 1,2,3) versus mild reactions (Arah8).

Study Population:

 Levels of peanut specific serum IgG4, with higher levels associated with increased tolerance to peanut protein.

Children ages 1-16 with peanut allergy suggested via history of reaction and objective evidence of IgE mediated hypersensitivity either via skin testing or in vitro testing (peanut specific IgE concentration) within the last 12 months.

### Inclusion criteria:

- Age 1-16 years
- History of immediate hypersensitivity reaction to peanut or a high level of suspicion based on testing at the discretion of the investigator
- Evidence of IgE mediated peanut hypersensitivity within a 12 month period of study enrollment including:
  - Skin prick test with wheal diameter of at least 3mm and/or
  - Peanut specific IgE >0.35 ku/L

### Exclusion criteria:

- History of life threatening peanut anaphylaxis
- Asthma requiring more than medium dose inhaled corticosteroids for age per the National Heart, Lung, and Blood Institute Asthma Guidelines
- Cardiovascular disease
- Use of beta-blockers (oral), angiotensin converting enzyme inhibitors, angiotensin receptor blockers, or calcium channel blockers
- Use of steroid medications in the following manners:
- Daily oral steroid dosing for greater than 1 month during the past year OR
- Burst or steroid course in the past 3 months before inclusion OR
- Greater than 2 burst oral steroid courses in the past year of at least 1 week duration
- Pregnancy or lactation
- Prior participation in food oral immunotherapy studies, including OIT, sublingual immunotherapy (SLIT), or epicutaenous immunotherapy (EPIT)
- Eosinophilic gastrointestinal disease
- Oat allergy, as oat flour is the vehicle with which study drug may be mixed for purposes of blinding and will be used as placebo for the exit DBPCFC

- History of food protein-induced enterocolitis syndrome (FPIES)
- History of developmental delay or speech delay that precludes age-appropriate communication, in the opinion of the investigator

Description of Sites and Facilities Enrolling Patients:

Screening will be performed at the Cleveland Clinic main campus and satellite outpatient clinic locations. Any patients identified as eligible will be referred to main campus for further evaluation and possible enrollment.

Description of Study Intervention:

Oral Immunotherapy will be administered utilizing a powder derived from boiled peanuts. Treatment will begin with an initial escalation day in which dosing is begun at 0.1 mg peanut protein and escalated to a final dose of 6 mg peanut protein. Doses are ingested orally. The subjects will continue daily oral ingestion of doses at home and return for updosing every 2 weeks to a final maintenance dose of 300 mg peanut protein. The subjects will continue daily oral ingestion of the peanut product for a minimum duration of 28 days before undergoing exit DBPCFC. At the conclusion of the study, patients will be offered continued maintenance therapy off study in line with current specialty standards.

Study Duration:
Participant Study Duration:

18 weeks 18 weeks

### 1.2 Study Schema



### 1.3 Schedule of Activities

| | l | | - 1 | | | ı | 1 | 1 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | | Study Visit 1 | Study Visit 2<br>Visit 1 +1-4 weeks | SV 3 Visit $2 + 2$ weeks | SV 4<br>Visit 2 +4 weeks | SV 5<br>Visit 2 +6 weeks | SV 6<br>Visit 2 +8 weeks | SV 7 Visit 2 +10 weeks | SV 8<br>Visit 2 +12 weeks | SV 9 Visit 2 +14 weeks | SV 10<br>Visit 1+18 weeks |
| Procedures | Enrollment/Baseline visit | Oral Food Challenge | Initial dose escalation | Dose escalation visit 1 | Dose Escalation Visit 2 | Dose escalation visit 3 | Dose escalation visit 4 | Dose escalation visit 5 | Dose escalation visit 6 | Dose escalation visit 7 | Oral Food Challenge |
| Informed<br>Consent | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Vitals | X | X | X | X | X | X | X | X | X | X | X |
| Spirometry* | X | | X | X | X | X | X | X | X | X | X |
| Blood Draw | | | X | | | | | | | | X |
| Skin prick test | | | X | | | | | | | | X |
| Oral food challenge | | X | | | | | | | | | X |
| Urine<br>Pregnancy | X | | | | | | | | | | X |
| Study Drug<br>Administration | | | X | X | X | X | X | X | X | X | |
| Study Drug<br>Compliance | | | | X | X | X | X | X | X | X | X |
| AE Review | | | X | X | X | X | X | X | X | X | X |
| Conmed<br>Assessment | X | X | X | X | X | X | X | X | X | X | X |

| FAQL | X | X |
|---------------|---|---|
| Questionnaire | | |

All dose escalation visits have a window of +/- 2 day

All follow up visits have a window of +/- 7 days

The enrollment/baseline visit, initial oral food challenge (SV 1), will take place at the Pediatric Allergy Clinic at the Cleveland Clinic main campus.

The initial escalation day, dose escalation visits, and final oral food challenge (SV 2-10) will take place in the Clinical Research Unit.

\* Spirometry will be performed on all patients ages 5+ and/or at the physician's discretion at the initial study visit as well as the exit oral food challenge. Rather than full spirometry, peak flow will be performed at every updosing visit on all patients ages 4+ and/or if the physician feels that it is developmentally appropriate

### 2. Introduction

### 2.1 Study Rationale

Peanut allergy (PA) is a common and potentially life threatening condition for which the only current approved management involves strict dietary avoidance. Oral immunotherapy (OIT) is a promising investigational treatment option for this condition, and multiple published studies have demonstrated efficacy in achieving successful desensitization to peanut in children with peanut allergy. 8-16 However, the widespread clinical use of OIT has been limited by numerous factors. These include the high rate of adverse events (AEs), including anaphylaxis, which often leads to high subject drop-out rates in published studies (Table 1). These studies all used peanut products produced by roasting methods, including flour, peanut powder, or peanut butter. Published data have demonstrated that boiling peanut results in reduced allergenicity while preserving the immunogenicity necessary to produce tolerance. 19 In this pilot study, we plan to compare the use of boiled peanut OIT to published data on roasted peanut OIT in children with peanut allergy. Based on currently available data, we hypothesize that the subjects treated with this novel regimen of boiled peanut will demonstrate lower rates of adverse events while demonstrating similar immunologic markers of peanut desensitization and possible tolerance compared to published data on subjects treated with OIT utilizing a traditional roasted peanut product.

### 2.2 Background and Significance

Peanut allergy (PA) has a reported prevalence of 2% in children and 0.7% in adults. The prevalence of PA also appears to be increasing, and in a registry of fatal food induced anaphylaxis, 63% of the 32 fatalities were caused by peanut. The implications of PA extend beyond the patient and their family. This food allergy in particular has impacted the educational system as well as the food industry. The effect on quality of life can be significant, foten leading to social isolation and even fear of death. Currently standard of care for PA consists of allergen avoidance, which is often ineffective, and administration of emergency medications on accidental exposure. Given the prevalence of PA and its associated morbidities, safe and effective therapies are desperately needed.

Immunotherapy relies on the delivery of increasing doses of specific allergens over time with the goal of developing desensitization, which increases the dose of protein needed to elicit an allergic response.

Over the past century, immunotherapy has been successfully used to treat asthma, allergic rhinitis, and insect venom anaphylaxis through subcutaneous or sublingual administration. Although the exact mechanisms underlying allergen immunotherapy are still not fully understood, it is known to induce allergen-specific regulatory T cells, which suppress TH2 responses that promote IgE production. This response is coupled with increases in serum concentrations of allergen-specific IgG4 antibodies which compete with IgE on cell surfaces and result in reductions in mast cell and basophil activation and mediator release. An increased IgG4 to IgE ratio is associated with clinical tolerance to a given food.

Though immunotherapy can be administered in a variety of methods, oral immunotherapy (OIT) has shown the most promise in the treatment of food allergy. Several recent trials have utilized the technique of oral immunotherapy for treatment of peanut and other food allergies. This therapy involves mixing the food allergen into a vehicle of choice and having the subject begin daily consumption while gradually increasing the dose. Several endpoints have been defined when evaluating the response to immunotherapy. Desensitization results in a higher threshold for an allergic reaction, typically above the amount that will be encountered in an accidental exposure. However, this does require ongoing dosing. The most desirable outcome of OIT is sustained unresponsiveness, or continued long term tolerance of the food without the need for daily maintenance therapy.

Although individual responses vary considerably, OIT will induce significant desensitization in most subjects who are able to tolerate the therapy. However, these studies are limited by frequent treatment related AEs and high rates of withdrawal due to these AEs. The reported AEs and dropout rates from representative studies are outlined in Table 1.8-16

There is a large amount of heterogeneity in the reporting of AEs. More specifically, AEs are at times reported in terms of the percent of subjects experiencing an adverse reaction. At other times, adverse reactions are reported in terms of the percent of doses that cause an AE. This method is often utilized to report AEs during maintenance dosing. This is in part due to the fact that over the course of all phases of an individual study and when including mild AEs in addition to more significant reactions, nearly 100% of patients have some form of AE during treatment. Thus it may be more meaningful to report the percent of doses causing symptoms at times.

Table 1: Prior OIT Trials

| Author | N | Age | Design | Adverse Events | Drop<br>outs | Additional Detail on Drop Outs |
|---|---|---|---|---|---|---|
| Jones et al<br>2009 [8] | 39 | 1-16 | Open label | 92% of subjects on initial escalation day, 46% doses during build up, 3.7% doses during maintenance | 10<br>(25%) | 4 withdrew for allergic effects and 6 for personal reasons |
| Hofmann<br>et al<br>2009 [10] | 28 | 1-16 | Open label | 93% of subjects on initial escalation day, 46% doses during build up, 3.5% of doses during maintenance | 5<br>(18%) | 3 withdrew following initial escalation, 1 during build up, 1 during maintenance |
| Blumchen<br>et al<br>2010 [9] | 23 | 3-14 | Randomized,<br>open label | 7.8% of doses during rush protocol, 2.9% of doses during maintenance | 8<br>(35%) | 1 during rush protocol, 7 during long term buildup of which 4 for allergic side effects |
| Varshney<br>et al<br>2011 [11] | 19 | 1-16 | Double blind,<br>placebo<br>controlled | 47% subjects with "clinically<br>relevant" AEs during initial<br>escalation day, 1.2% doses during<br>build up | 3<br>(16%) | 2 withdrew during initial escalation day and 1 after first build up dose |
| Anagnostou<br>et al | 22 | 4-18 | Open label | 86% subjects during build up and maintenance | 1<br>(5%) | Withdrew after the first up dose at home |

| | | | | | | - |
|---|---|---|---|---|---|---|
| 2011 [12] | | | | | | |
| Anagnostou<br>et al<br>2014 [13] | 99 | 7-16 | Randomized,<br>placebo<br>controlled<br>cross over | 6.3 % of all doses | 7<br>(7%) | 5 withdrew for allergic reactions or persistent symptoms, 1 disliked taste, and 1 no specific reason |
| Vickery et al 2014 [14] | 39 | 1-16 | Open label | Previously reported in pilot study (Jones et al 2009) | 15<br>(38%) | 6 withdrew due to allergic side effect and 9 for personal reasons |
| Narisety et<br>al<br>2014 [15] | 21 | 7-13 | Randomized,<br>double blind,<br>placebo<br>controlled | 43% doses during blinded phase (escalation and maintenance), 36.7% doses in OIT group during unblended phase | 7<br>(33%) | 1 withdrew after initial escalation,<br>1 during build up and 3 during<br>maintenance. 1 drop out on SLIT<br>with placebo OIT |
| Vickery et al<br>2016 [16] | 37 | 9-36<br>months | Randomized,<br>double blind,<br>low and high<br>dose | 95% patients during entire study,<br>0.8% doses during study | 5<br>(14%) | 2 withdrew for nonadherence, 1 for recurrent emesis and 1 for EoE |

Abbreviations: N, number of subjects, AEs, adverse events, SLIT, sublingual immunotherapy, OIT, oral immunotherapy, EoE, eosinophilic esophagitis

Given the high rate of these treatment related AEs such as oral itching, stomach upset and other GI complaints, and occasional serious systemic allergic reactions requiring the use of injectable epinephrine, OIT is still considered an experimental treatment. While some major medical centers and a number of private practice allergists offer peanut OIT to their patients, it is not yet FDA approved.

A commercially developed product, AR101 (Aimmune Therapeutics), an investigational oral biologic drug, was recently trialed in a phase 3 study evaluating efficacy. In the intervention group, 67.2% of patients ages 4-17 tolerated at least a 600-mg dose of peanut protein in the exit food challenge, compared to 4.0% of placebo patients (p<0.00001). In the trial's primary analysis group of ages 4-17, 496 patients from both arms (372 AR101 and 124 placebo) were evaluable for safety. In both arms, the incidence of serious adverse events (SAEs) was low. A total of 10 patients experienced SAEs, none of which were considered life-threatening: nine of these patients were in the AR101 arm (2.4%) and one was in the placebo arm (0.8%). Of the nine AR101 patients who experienced a SAE, five patients experienced mild or moderate SAEs. The other four AR101 patients experienced severe SAEs, which, for two of these patients, were not related to treatment (a concussion and a viral asthmatic exacerbation). Of the two patients who experienced severe SAEs related to treatment, both of whom had elevated baseline peanut-specific IgE levels greater than 100 kU/L, one experienced anaphylaxis, and the other experienced wheezing on the first day of treatment. Both of these patients discontinued from the study. In ages 4–17, 20.4% of AR101 patients and 6.5% of placebo patients discontinued the trial. In the AR101 arm, 12.4% of patients discontinued due to investigator-reported adverse events, including 6.7% due to gastrointestinal adverse events and 2.7% due to systemic allergic hypersensitivity reactions. In the placebo arm, 2.4% of patients discontinued due to investigator-reported adverse events (Table 2).<sup>28</sup>

Table 2: Discontinuations in the AR101 Group<sup>28</sup>

| | | 101<br>372) |
|---|---|---|
| | % | n |
| Total discontinuations regardless of causality | 20.4% | 76 |
| Discontinuations not related to adverse events | 8.0% | 30 |
| Discontinuations related to adverse events | 12.4% | 46 |
| Gastrointestinal <sup>2</sup> | 6.7% | 25 |
| <ul> <li>Systemic hypersensitivity reactions<sup>3</sup></li> </ul> | 2.7% | 10 |
| Respiratory system | 1.1% | 4 |
| Cutaneous | 0.8% | 3 |
| Other | 1.1% | 4 |

We seek to identify a means of accomplishing peanut desensitization while decreasing the rate of treatment related AEs. It has been shown that standard roasting methods of peanut preparation can play a significant role in increasing the undesirable allergenic properties of peanuts.<sup>17</sup> It has also been demonstrated that peanut antigen stimulation of peripheral blood T lymphocytes is unaffected by various heating methods, which is necessary for induction of tolerance.<sup>18</sup> An additional study confirms the findings of extended boiling resulting in reduction of peanut allergenicity while preserving the effect on T cell reactivity.<sup>19</sup> A group recently reported a series of 4 subjects with peanut allergy who were treated with daily doses of boiled peanut, one of which subsequently transitioned to raw peanut. All subjects demonstrated lower IgE reactivity to boiled peanut compared to control suggesting that in vivo findings correlate with the prior in vitro data.<sup>20</sup>

While OIT is a promising therapy, we hypothesize that by treating peanut allergic subjects with a peanut product of reduced allergenicity but preserved T cell reactivity, we will be able to desensitize these subjects to a target maintenance dose of peanut protein with reduced rates of allergen associated AEs, while preserving immunologic effects that will promote tolerance. This will confirm that the immunologic changes produced by roasted peanut OIT can be replicated more safely using boiled peanut. If successful, such a therapy will decrease the number of subjects that must discontinue this treatment due to related AEs, and offer a potentially important therapy for this life threatening condition. Improved safety of this intervention may also allow for higher treatment doses to be used, may allow inclusion of more severely allergic subjects excluded from previous trials, and possibly increase the likelihood for attainment of permanent tolerance with sustained unresponsiveness, rather than perpetuating the need for continual daily dosing. This will likely result in the eventual inclusion of BPOIT in general Allergy/Immunology practice as a treatment for peanut allergy. We suspect this therapy will improve quality of life as measured by validated questionnaires as well as, or better than, roasted peanut oral immunotherapy.<sup>28</sup>

### 2.3 Risk/Benefit Assessment

### 2.3.1 Known potential risks

There is a significant rate of adverse reactions with peanut oral immunotherapy in clinical trials to date. Mild adverse reactions such as oral itching or nausea are reported in up to 10-15% of all doses. Over the course of an individual study, this reaches nearly 100% of all subjects. The rate of these adverse events are outlined in representative studies in Table 1.

More severe reactions requiring treatment with epinephrine or inhaled beta-agonists are less frequent but can occur. In a large review of multiple centers performing peanut OIT, Wasserman et al noted a total of 95 adverse reactions requiring epinephrine in 352 patients that collectively received more than 240,000 doses of peanut.<sup>25</sup> The results of the largest peanut OIT trial to date, a phase 2 clinical trial utilizing product AR101 were published in March of 2018.<sup>21</sup> In this study, 9 (14%) of 63 subjects received a single injection of epinephrine during initial double blind placebo controlled food challenge (DBPCFC) at screening: 4 were randomized to AR101, 4 to placebo, and 1 was not enrolled. For the duration of maintenance therapy, one treatment subject received a single epinephrine injection for moderate anaphylaxis at home. Finally, during the exit DBPCFC, 11 of 26 placebo subjects (42%) were administered epinephrine and 2 of 23 AR101 subjects (9%) received a single injection of epinephrine.

Across the various peanut OIT trials, there has been no specific statistical analysis examining adverse reaction rate or withdrawal rate at various ages. Presumably this is due to the fact that no specific age related pattern has emerged and that anaphylaxis and subject withdrawal has occurred in subjects of all ages.

There is also a risk for development of Eosinophilic Esophagitis (EoE). A recent review estimated the prevalence across the OIT clinical trials as 3-4% and in the study conducted by Bird et al, EoE occurred in only 1 subject (<5%) from the treatment group.<sup>21</sup> Once OIT is discontinued in these patients, the EoE typically resolves.

There is also a risk of causing anxiety or stress in the subject or the family. The impact of oral immunotherapy on quality of life has been examined with a variety of foods. Quality of life in patients with food allergy improves in some but declines in others while undergoing OIT, and in particular tends to decline in those rating a higher quality of life prior to initiation of the treatment.<sup>26</sup>

### 2.3.1 Known Benefits

The primary benefit of peanut oral immunotherapy is increasing the threshold of peanut which will result in an allergic reaction. This increased threshold is typically above the amount encountered upon accidental ingestion. This can reduce the risk of a subject experiencing a severe or life-threatening allergic reaction due to an accidental ingestion. Importantly, this can also ease anxiety in both the subject and family that is often associated with the diagnosis of a food allergy.

The question of whether oral immunotherapy will induce sustained unresponsiveness, or ongoing tolerance of peanut following cessation of the daily maintenance doses, is yet to be fully elucidated.

Results have varied among initial clinical trials. If this can be obtained, this would allow full incorporation of peanut into the diet of previously allergic subjects.

### 2.3.3 Assessment of the potential risks and benefits

We believe that given the low rate of serious adverse reactions along with the hypothesis that subjects receiving the boiled peanut will experience a lower rate of these adverse reactions, that the potential benefit to induce desensitization to peanut outweighs these risks. In addition to personal benefit, this study has the potential to further the future treatment options for peanut allergic children.

### 3. Objectives and Endpoints

| Objective | Endpoints | Justification |
|---|---|---|
| Primary | | |
| Determine the effect of boiled peanut immunotherapy on the immune response to peanut and demonstrate that the proportion of subjects successfully desensitized with boiled peanut OIT is not appreciably lower than the proportion of subjects successfully desensitized with roasted peanut OIT in published data. | Primary Endpoint: Response to treatment defined as ability to successfully consume a single dose of 300 mg or greater of peanut protein with no dose limiting symptoms at exit double blind placebo controlled food challenge (DBPCFC). The highest dose of roasted peanut protein tolerated by the subject at exit DBPCFC will also be compared to the highest dose tolerated at baseline. | Previous in vitro data has demonstrated that boiling peanuts can result in reduction of peanut allergenicity while preserving the effect on T cell reactivity. |
| | The effect of boiled peanut immunotherapy on the immune response to peanut will be evaluated via specific serum markers of sensitization and tolerance to peanut. • Levels of serum specific peanut IgE, with higher levels associated with greater likelihood of clinical reaction on exposure to peanut protein. • Peanut protein component panel, to determine the presence of high levels of sensitivity to peanut proteins known to be | |

- associated with severe systemic reactions (Arah 1,2, 3) versus mild reactions (Arah8)
- Levels of peanut specific serum IgG4, with higher levels associated with increased tolerance to peanut protein
- These markers will be evaluated at baseline and the conclusion of the study.

### Secondary

Compare the rate of adverse effects of boiled peanut oral immunotherapy to published data on roasted peanut oral immunotherapy.

The rate of adverse events in the subjects receiving boiled peanut oral immunotherapy. Possible adverse events include: side effects of treatment defined as oral itching, rhinorrhea, conjunctivitis, urticaria, angioedema, abdominal upset, vomiting, diarrhea, cough, wheeze, or anaphylaxis

- Adverse events will be recorded in terms of the percentage of subjects with adverse events on initial escalation day and at dose escalation visits by CRU staff.
- Adverse events will also be recorded in terms of overall percentage of home doses that result in adverse reaction, with data compiled from home logs (Supplement 2).

The adverse reactions will be graded in severity and the treatment required will be recorded.

Validated, age-specific, foodrelated quality-of-life surveys before and after peanut oral immunotherapy will be completed As described above, the rate of adverse events with roasted peanut oral immunotherapy is high. Thus treatment options with less adverse effects are highly desirable. In vitro data has demonstrated that boiled peanut has reduced allergenicity compared to roasted peanut and similar immunogenicity. As such, we anticipate a lower rate of adverse reactions in our subjects compared to published data on roasted peanut OIT.

| by all patients/families <sup>27</sup> |
|----------------------------------------|
| (Supplement 1). |

### 4. Study Design

### 4.1 Overall Design

We will perform a phase 1 clinical trial utilizing oral immunotherapy with powder derived from boiled peanut. Our hypothesis is that the subjects treated with this novel regimen of boiled peanut will demonstrate lower rates of adverse effects while demonstrating similar immunologic markers of peanut desensitization and possible tolerance in comparison to published data on subjects treated with OIT utilizing roasted peanut product.

### 4.2 Scientific Rationale

Oral immunotherapy has not yet been approved by the FDA for the treatment of food allergy. However, multiple clinical trials in recent years have shown significant promise in utilizing oral immunotherapy for peanut allergy. It is expected that oral immunotherapy will be more widely available in the near future, and options with a more favorable side effect profile are highly desirable.

The phases of our clinical trial were modeled after the previous high quality studies utilizing roasted peanut OIT and are comparable in methodology and duration.

### **4.3 Justification for Dose**

The maintenance dose for oral immunotherapy with peanut has varied across previous clinical trials. Doses have ranged from 300 mg up to a maximum of 4000 mg.<sup>8-16</sup> Only one study has compared the efficacy of different maintenance doses. In this study, Vickery et al found that a maintenance dose of 300 mg was as efficacious as a 3000 mg dose at inducing sustained unresponsiveness. This is also likely to be above the dose encountered in an accidental ingestion, as 1 whole peanut contains roughly 250 mg of peanut protein.<sup>22</sup>

### 4.4 End of Study Definition

A participant is considered to have completed the study if he or she has completed all phases of the study including the last visit or the last scheduled procedure shown in the Schedule of Activities (SoA), Section 1.3.

The end of the study is defined as completion of the last visit or procedure shown in the SoA.

### 5. Study Population

We will recruit 10 children ages 1 to 16 years with peanut allergy suggested via history and objective evidence of IgE mediated hypersensitivity to peanut either via skin testing or in vitro testing (peanut specific IgE concentration) within the last 12 months. Skin prick testing will be performed with standard peanut extract (1:20 w/v, Greer) and peanut specific IgE concentration will be performed using ImmunoCap. We will use standard criteria to indicate sensitization.

### 5.1 Inclusion Criteria

#### **Inclusion Criteria**

Age 1-16 years

History of immediate hypersensitivity reaction to peanut or a high level of suspicion based on testing at the discretion of the investigator

Evidence of IgE mediated peanut hypersensitivity within a 12 month period of study enrollment

SPT with wheal/flare of at least 3 x 6 mm and/or
Peanut specific IgE >0.35 kU/L

Abbreviations: SPT, skin prick test

In addition, the individual's parent or guardian must provide signed and dated informed consent and the individual must provide signed and dated assent when appropriate. The individual and parent or guardian must agree to comply with all study procedures and the individual must have the ability to take oral medication.

### 5.2 Exclusion Criteria

### **Exclusion Criteria**

History of life threatening peanut anaphylaxis

Asthma requiring more than medium dose ICS

Prior participation in OIT, SLIT or EPIT

Oat allergy

**Cardiovascular Disease** 

Use of beta-blockers (oral), angiotensin converting enzyme inhibitors, angiotensin receptor blockers, or calcium channel blockers

Use of steroid medications in the following manners:

Daily oral steroid dosing for greater than 1 month during the past year OR Burst or steroid course in the past 3 month before inclusion OR

Greater than 2 bursts oral steroid courses in the past year of at least 1 week duration

### **Pregnancy or lactation**

### **Eosinophilic Gastrointestinal Disease**

History of food protein-induced enterocolitis (FPIES)

History of developmental delay or speech delay that precludes age-appropriate communication, in the opinion of the investigator

Abbreviations: ICS, inhaled corticosteroid, OIT, oral immunotherapy, SLIT, sublingual immunotherapy, EPIT, epicutaneous immunotherapy

A history of life-threatening anaphylaxis is defined as a reaction involving respiratory failure, hypotension or neurologic compromise. Medium dose ICS is defined by the National Heart, Lung, and Blood Institute asthma guidelines. Patients with oat allergy, while rare, are to be excluded as this will serve as the placebo for our exit food challenge (SV10).

### **5.3 Lifestyle Considerations**

With the exception of the oral immunotherapy treatment, subjects will be instructed to continue strictly avoiding peanut in their diet. Prior oral immunotherapy studies have sought to determine predictors of adverse reactions to treatment and co-factors are often noted in subjects that do experience adverse reactions. This can include illness, exercise, or allergen exposure in subjects with allergic rhinitis. Subjects will be instructed to refrain from exercising for 60 minutes following ingestion of the study drug. Subjects and their families will also be instructed to contact the physician investigators if an illness or significant rhinitis symptoms occur, as a temporary adjustment to the daily dose may be necessary.

### **5.4 Screen Failures**

Screen failures are defined as participants who consent to participate in the clinical trial but are not subsequently randomly assigned to the study intervention or entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants, to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any serious adverse event (SAE).

Individuals who do not meet the criteria for participation in this trial (screen failure) because there are no objective signs of an IgE mediated reaction during initial food challenge may not be rescreened. These individuals are not peanut allergic and thus not candidates for the treatment of peanut allergy.

### 5.5 Strategies for Recruitment and Retention

Individuals will be screened for possible study eligibility at the Cleveland Clinic Allergy Clinic locations. The recruiting physicians will include the Pediatric Allergy clinic staff as well the Respiratory Institute Allergy staff. All Allergy physicians will be made aware of the study and details of recruitment at a Quarterly Allergy and Immunology staff meeting which is attended by both Pediatric Institute and Respiratory Institute allergy physicians.

Once potential participants are identified, a study investigator will reach out to the parent/guardian of the patient via an introductory letters and telephone to inquire about study interest. Should the family express a desire to participate, they will be invited to the main campus for Enrollment/Baseline visit. This visit will take place with one of the physician investigators and will involve extensive discussion of the study including protocol, risks and benefits. If the individual and their parent or guardian opt to participate in the study, informed consent, and assent when appropriate, will be obtained at this time and the individual will be enrolled.

There has been a significant amount of media and online attention to these evolving treatment options for food allergy including OIT. As such, frequent and unsolicited inquiries regarding OIT are made by patients/families encountered in the Allergy clinics. This fact accompanied by the prevalence of peanut allergy in the pediatric population leads us to believe the accrual rate of participants will be fairly rapid.

### 6. Study Intervention

### **6.1 Study Interventions Administration**

### 6.1.1 Study Intervention Description

Commercially available whole canned boiled peanuts (Peanut Patch, McCall Farms) will be purchased from online retailers. This commercially available product, regulated by the Food and Drug Administration, is regularly consumed by humans.

Although additives are typically contained in commercially available products, this is not expected to be clinically relevant. The prevalence of allergy to food additives has been reported as high as 0.23% based on self-report. However, the reported cases in medical literature are typically either anecdotal or diagnosed based on poorly-controlled challenge procedures. Thus expert consensus is that relatively few food additives have been convincingly demonstrated to true hypersensitivity reactions.<sup>6</sup>

### **Peanut Patch**

Information from the Manufacturer's Website:

### **Nutrition Facts**

Serving Size 1/4 cup (about 34g)

**Amount Per Serving** 

Calories 100Calories from Fat 70

| | % Daily | Value* |
|--------------------|--------------|--------|
| Total Fat 8g | | 12% |
| Saturated Fat 1.5g | | 8% |
| Trans Fat 0g | | |
| Cholesterol 0mg | | 0% |
| Sodium 320mg | | 13% |
| Total Carbohydrate | <b>9</b> 3g | 1% |
| Dietary Fiber 2g | | 8% |
| Sugars 0g | | |
| Protein 4g | | |
| Vitamin A 0% | Vitamin C 0% | |
| Calcium 0% | Iron 2% | |

<sup>\*</sup> Percent Daily Values are based on a 2,000 calorie diet. Your daily values may be higher or lower depending on your calorie needs:

### Calories per gram:

Fat 9 • Carbohydrate 4 • Protein 4

The boiled peanuts will be processed into powder. All processing will take place in the University Hospitals Dahms Clinical Research Unit kitchen. The Dahms Clinical Research Unit kitchen is a Class III Non-Commercial Food Service establishment and is inspected on a routine basis through the Cleveland Health Department. The peanut processing will be supervised by the CRU Bionutrition director who is certified in food protection through the Ohio Department of Health.

Boiled peanuts will be shelled and placed evenly on individual trays of a food dehydrator purchased for use of this process only (Nesco FD-75a Food Dehydrator). The dehydrator was purchased specifically for this study and no other food items will come into contact with or be used on this device. Peanuts will be dehydrated at a temperature of 105 degrees F (41 degrees C) for 17 hours (1,020 minutes). Immediately upon removal, peanuts will be ground to a fine powder in a food processor.

Peanut powder will be placed in Pactiv/Newspring plastic deli containers with lids. These will be sealed, labeled, and shipped via courier from the Case Western Clinical Research Unit directly to the investigational drug pharmacy for storage in a refrigerator.

We will characterize the processed boiled peanut and determine the concentration of peanut protein. This will be necessary to calculate the doses for subjects in the boiled peanut immunotherapy arm. To further characterize this product, the specific component proteins including Ara h 1, 2, 3, 8 and 9 will also be quantified. These specific proteins are known to be associated with either higher risk for anaphylaxis (Ara h 1, 2, and 3) versus more mild reactions (Ara h 8).24 This assay will be performed as an ELISA within the Cleveland Clinic Proteomics lab.

A representative sample from each batch of prepared boiled peanut powder will be sent to JLA laboratories, a USDA certified lab, in order to test for aflatoxin levels and to quantify a total bacterial count and total mold count. This lab is approved by the USDA-AMS for Aflatoxin in Peanuts and ISO 17025 accredited by ANAB for aflatoxin and microbiological testing. Aflatoxin testing is performed by HLPC method in accordance with AOAC 991.31 and AOAC 2005.08. The total bacterial count will be obtained using AOAC-RI 051702/MB073.6 and the mold count using AOAC-RI 051702/MB074.03.

The doses will be measured and allotted into individual medicine cups by the Investigational Drug Service Department as outlined in Section 6.2. The subjects will mix the powder with a vehicle of the subject/family's choice (applesauce, pudding, or hot cereal) just prior to oral ingestion.

### 6.1.2 Dosing and Administration

### Oral Food Challenge

After informed consent is obtained (and assent when relevant), eligible subjects will undergo an open roasted peanut graded food challenge to 4000 mg of peanut protein to confirm peanut allergy and to determine the amount of peanut protein required to induce an allergic reaction at baseline. An oral food challenge is the gold standard for diagnosis of food allergy. PB2 peanut powder (PB2 Foods, Tifton, GA) will be used exclusively for this challenge, mixed in a vehicle of the family's choice (such as applesauce, pudding, etc).

Subjects will be instructed to hold medications with strong antihistamine properties for five days prior to the challenge (diphenhydramine, loratadine, desloratadine, cetirizine, levocetirizine, fexofenadine, azelastine). The challenge will not be performed in the setting of acute illness, including febrile illness, asthma exacerbations, and significant flares of atopic dermatitis.

The oral food challenge protocol is outlined in Table 3. The initial oral food challenge will take place under the supervision of a trained Allergy/Immunology investigator and trained Allergy/Immunology nurse at Cleveland Clinic Children's main campus Allergy Clinic, where similar food challenges are routinely conducted. The physician investigator available will be trained in recognition and treatment of IgE mediated food reactions, will be available for immediate evaluation of any signs or symptoms of reaction.

Table 3: Oral food challenge to peanut for enrollment (Study Visit 1)

| | 1_ | 1 |
|---|---|---|
| Time | Dose | Clinician Intervention * |
| 0 | 5mg | Obtain weight, temperature, heart rate, blood pressure, |
| | | respiratory rate, and oxygen saturation level. Peak flow will |
| | | be done on patients 4+ or deemed developmentally |
| | | appropriate. Full physical examination of ears, oropharynx |
| | | and nose, lungs, and skin prior to administration of dose |
| +15 minutes | 10mg | Examination of skin and auscultation of lungs prior to dose |
| +30 minutes | 25mg | Examination of skin and auscultation of lungs prior to dose |
| +45 minutes | 50mg | Examination of skin and auscultation of lungs prior to dose |
| +60 minutes | 100mg | Examination of skin and auscultation of lungs prior to dose |
| +75 minutes | 500mg | Examination of skin and auscultation of lungs prior to dose |
| +90 minutes | 1000mg | Examination of skin and auscultation of lungs prior to dose |
| +105 minutes | 4000mg | Examination of skin and auscultation of lungs prior to dose |
| | | Full physical examination of ears, oropharynx and nose, |
| | | lungs, and skin after completion of final dose. |
| | • | |

<sup>\*</sup>Vital signs including heart rate, blood pressure, respiratory rate and oxygen saturation level to be obtained with any change in physical exam or clinical status

If objective signs of an allergic reaction occur, then the challenge will be stopped, and the subject treated based on the presenting symptoms and clinical judgment of the supervising investigator (Table 4). If no objective signs occur within 2 hours after the last dose is consumed, then the child will be considered not peanut allergic and will not qualify for the study.

### Table 4: Oral food challenge stopping criteria

A positive food challenge will be defined by the presence of either of the following:

- One or more major criteria
- Two or more minor criteria

An indeterminate food challenge will be defined by the presence of one minor criterion.

A negative food challenge will be defined by the absence of major or minor criteria.

All symptoms should be of new onset and not due to ongoing disease. Symptoms must occur no later than 2 hours after the last dose.

### Major Criteria

- Confluent erythematous pruritic rash
- Respiratory signs (at least one of the following):

Wheezing

Inability to speak

Stridor

Dysphonia

**Aphonia** 

- >/= 3 noncontact urticarial lesions lasting for more than 3 minutes
- >/= 1 site of angioedema
- Hypotension for age not associated with vasovagal episode
- Evidence of severe abdominal pain (such as abnormal stillness or doubling over) that persists for more than 3 minutes

### Minor Criteria

- Vomiting (persistent symptoms would elevate to major criterion)
- Diarrhea
- Persistent rubbing of nose or eyes that lasts for >/= 3 minutes
- Persistent rhinorrhea that lasts for >/= 3 minutes
- Persistent scratching that lasts for >/= 3 minutes

The subjects with objective signs of an IgE mediated reaction to peanut using standard criteria (Table 4) will be eligible for enrollment.

If patient is found to be study eligible, then a urine pregnancy test will be done on females who have reached the age of child birthing potential.

### **Initial Dose Escalation**

Upon enrollment, demographic data will be collected including age, sex, race, history of asthma/atopic dermatitis/allergic rhinitis. The enrolled subjects will present to the Clinical Research Unit for a one day dose escalation. The intent of the initial escalation is to begin and remain at subthreshold levels and identify a safe starting dose for home administration. Any subjects unable to tolerate at least 1.5 mg peanut protein will be discharged.

Active illness or asthma exacerbation will prompt rescheduling of the initial dose escalation. Patients are encouraged to eat foods brought from home before and during dose escalation.

Prior to the first dose, patients will receive the following interventions:

- Blood obtained by venipuncture for baseline laboratory evaluation
  - Peanut specific IgE concentration
  - Peanut component testing (peanut specific IgE concentration for Ara h 1, 2, 3, 8 and 9)
  - o Peanut specific IgG4 concentration.
  - Serum samples will be sent to the Cleveland Clinic Main Campus laboratory with the exception of the peanut IgG4 level which will be sent out to the Mayo Clinic.
- Skin prick test to peanut with extracts routinely used for this purpose in clinical practice
  - Negative control (50% glycerin/50%Cocas)
  - Positive control (Histamine base 6mg/mL)
  - Peanut extract 1:20 (Hollister Stier)
  - Apply one drop of each solution to upper back (infants and young children) or forearm (children over the age of 6 able to avoid scratching the extract), and prick through with sterile bifurcated needle to disrupt the top layer of the epidermis. The location used for the skin prick test will remain consistent for each patient throughout the study.
  - The test will be read by the clinician 15 minutes following application. The wheal (raised center) and flare (flat erythematous patch) will be measured horizontally and vertically with an average of these 2 measurements recorded as the diameter.

Table 5: Initial dose escalation (Study Visit 2)

| Time | Dose | Clinician Intervention * |
|---|---|---|
| 0 | 0.5 mg peanut | Obtain weight, temperature, heart rate, blood pressure, |
| | protein | respiratory rate, and oxygen saturation level (i.e. vital signs). Peak |
| | | flow will be measure on patient 4+ or deemed developmentally |
| | | appropriate. Full physical examination of ears, oropharynx and |
| | | nose, lungs, and skin prior to administration of dose |
| +30 minutes | 1 mg | Repeat vital signs. Examination of skin and auscultation of lungs |
| | | prior to dose |
| +60 minutes | 2 mg | Repeat vital signs. Examination of skin and auscultation of lungs |
| | | prior to dose |
| +90 minutes | 4 mg | Repeat vital signs. Examination of skin and auscultation of lungs |
| | | prior to dose |
| +120 minutes | 6 mg | Repeat vital signs. Examination of skin and auscultation of lungs |
| | | prior to dose |

<sup>\*</sup>Vital signs including heart rate, blood pressure, respiratory rate and oxygen saturation level to be obtained with any change in physical exam or clinical status

Dose escalation will begin with 0.5 mg of peanut protein and increase to a maximum of 6 mg (Table 5). The doses will be administered at 30 minute intervals following a set of vital signs and limited physical examination. At any objective sign of reaction (Table 4) the escalation will stopped, and the patient will be treated based on the presenting symptoms and clinical judgment of the supervising investigator. Subjects will be monitored for 2 hours after resolution of any signs of reaction and/or after completion of the final dose.

Subjects will then be instructed to consume the highest tolerated dose of peanut protein daily until their return for dose escalation.

### Build-Up

For the next phase, participants will undergo incremental dose escalations every two weeks. These dose escalations with take place under the supervision of a trained Allergy/Immunology physician investigator within the Clinical Research Unit. The subject will be given an increased dose of the peanut and observed for at least 2 hours. Subjects will then continue to take daily doses of an identical amount of peanut protein at home. We will increase to a target maintenance dose of 300 mg of peanut protein, which should be accomplished in approximately 6 dose increases, or 12 weeks' time.

If a patient is unable to tolerate the maximum dose during the initial dose escalation visit, they will be given double the maximum dose tolerated during the dose escalation visits until they are back on the dose escalation schedule defined in Table 6.

If a subject does not tolerate a dose increase, then the patient will be administered a dose reduced by 25%, with increase to the originally intended dose at the subsequent visit. If the patient still does not tolerate the dose, then the decision on how to proceed will be determined at the investigator's discretion. This may involve temporarily decreasing the subject's dose, making a smaller increase, or prolonging the duration of a given dose. If any subject is unable to reach the goal maintenance dose, then the investigator may decide to continue the subject on a lower maintenance dose for the duration of the study.

**Table 6: Dose Escalation Schedule** 

| Dose of Peanut Protein | Week of Protocol |
|------------------------|------------------|
| 6 mg | 0 |
| 12 mg | 2 |
| 25 mg | 4 |
| 50 mg | 6 |
| 75 mg | 8 |
| 150 mg | 10 |
| 300 mg | 12 |

### **Home Dosing**

All subjects will be offered the opportunity to continue once daily consumption of the maintenance dose after the end of their study participation. This ongoing maintenance therapy is optional and will not be paid for by the study. The subjects will be instructed to otherwise continue a peanut free diet.

### Follow Up

The subject will also undergo a final oral food challenge at the final visit (SV10). This food challenge will be double blind and placebo controlled. A double blind placebo controlled food challenge (DBPCFC) is the gold standard for diagnosis of food allergy and is the standard utilized for most oral immunotherapy trials at exit.

Roasted peanut powder will be utilized for the challenge, with oat flour as placebo. An individual will undergo a standard challenge described below (Table 7) with either the roasted peanut or the placebo, blinded to both subject and investigators. The same individual will then undergo a second challenge with the opposite (either peanut or placebo) either later that day or by returning to clinic the following day. Each challenge will be performed by increasing doses up to a final dose of 1000 mg of peanut protein. The individual doses will be 25, 100, 200, 300, 600, and 1000 mg of peanut protein. The highest tolerated dose will be recorded. If a patient reacted to a dose lower than 25 mg of peanut powder during the initial Oral Food Challenge then they will be started at the dose lower than where the reaction occurred for the DBOFC.

A urine pregnancy test will be repeated on all females of child bearing potential before the DBOFC.

Table 7: Double blind oral food challenge to peanut or control oat (SV 10)

| Time | Dose | Clinician Intervention * |
|---|---|---|
| 0 | 25 mg peanut<br>protein | Obtain weight, temperature, heart rate, blood pressure, respiratory rate, and oxygen saturation level. Peak flow in children ages 4+ or as developmentally appropriate. Full physical examination of ears, oropharynx and nose, lungs, |
| L1E minutos | 100 mg | and skin prior to administration of dose |
| +15 minutes | 100 mg | Examination of skin and auscultation of lungs prior to dose |
| +30 minutes | 200 mg | Examination of skin and auscultation of lungs prior to dose |
| +45 minutes | 300 mg | Examination of skin and auscultation of lungs prior to dose |
| +60 minutes | 600 mg | Examination of skin and auscultation of lungs prior to dose |
| +75 minutes | 1000 mg | Examination of skin and auscultation of lungs prior to dose |
| | | Full physical examination of ears, oropharynx and nose, |
| | | lungs, and skin after completion of final dose. |

<sup>\*</sup>Vital signs including heart rate, blood pressure, respiratory rate and oxygen saturation level to be obtained with any change in physical exam or clinical status

If objective signs of an allergic reaction occur, then the challenge will be stopped, and the subject treated based on the presenting symptoms and clinical judgment of the supervising investigator (Table 4). If no objective signs occur within 2 hours after the last dose is consumed, then the challenge will be considered negative.

### Quality of Life Questionnaire

At enrollment and after completion of the study, patients or caregivers will be asked to complete previously validated, age specific food allergy quality of life questionnaires<sup>27</sup>( **Supplement 1**)

### **6.2 Preparation/Handling/Storage/Accountability**

The Investigational Drug Service (IDS) will provide secure storage, temperature monitoring, drug accountability, and dispensing of Investigational Product (IP) to comply with the protocol and applicable state and federal regulations related to clinical research.

### **IP Management**

Upon the receipt of the IP, IDS will electronically document lot numbers, expiration dates, and quantity. The supply of roasted peanut powder and boiled peanut powder will be tracked and stored separately.

### IP dispensing

IDS will dispense the IP to eligible subjects upon receipt of a valid prescription. The prescription will be scanned to <a href="mailto:ids@ccf.org">ids@ccf.org</a> or faxed to 216 445-5554, Monday through Friday, 0700-1600. After reviewing the prescription, the pharmacist will:

- 1. Weigh the prescribed dose
- Transfer the prescribed dose into a plastic jar
- 3. Dispense the quantity of doses prescribed
- 4. Update drug accountability log\*\*
- 5. File the prescription in the subjects' tab in the study binder

### IP disposition

Returned or expired IP will be accounted for and then destroyed per department policy.

### 6.3 Measures to Minimize Bias

This study utilizes a prospective trial design in order to minimize recall bias. In addition, the double blind placebo controlled exit challenge will help minimize bias.

### **6.4 Study Intervention Compliance**

The subjects will have periodically scheduled trips to return the empty medicine cups for monitoring of adherence. In addition, the subjects or their families will complete a log at home recording administration of doses as well as any adverse effects.

### **6.5 Concomitant Therapy**

Data regarding the subjects' concomitant medications will be recorded at each study visit to the Pediatric Allergy Clinic or the Clinical Research Unit. For this protocol, a prescription medication is defined as a medication that can be prescribed only by a properly authorized/licensed clinician. Medications to be reported include concomitant prescription medications, over-the-counter medications such as oral antihistamines, and supplements.

The concomitant use of antihistamines could directly affect the primary endpoint. The use of antihistamines could mask or prevent some symptoms of an allergic reaction such as urticaria or pruritus. Upon enrollment, the treating physician investigator will evaluate the specific indication for antihistamine use and will make a determination regarding continued use or discontinuation. This will be documented within the electronic medical record.

<sup>\*\*</sup> Associate the dose, quantity, lot of IP dispensed with subject number and date

### 6.5.1 Rescue Medication

All subjects will be prescribed an epinephrine auto-injector to have available for rescue at home. All subjects will also be prescribed an oral antihistamine, cetirizine, to have available for rescue at home. It will be confirmed that all subjects with an underlying diagnosis of asthma have a prescription for a short acting beta-agonist (albuterol or levalbuterol) available for rescue at home. Any subjects with a diagnosis of asthma that do not have a short acting beta-agonist will have one prescribed.

The study sites (Pediatric Allergy office and Clinical Research Unit) will have rescue medications available at the time of each study visit. The following rescue medications may be used:

| Treatment | Adult Dose | Route | Dosing Interval | Special Considerations | Pediatric Dose |
|---|---|---|---|---|---|
| EPINEPHRINE<br>IM/SQ | 1:1000 concentration<br>0.3mg (range 0.3-<br>0.5mg, maximum<br>1mg per dose) | IM vastus lateralis<br>(lateral thigh) is<br>recommended site<br>for quickest<br>absorption.<br>Can also be given<br>SQ or IM in<br>deltoid. | Every 5 to 10<br>minutes prn<br>or sooner if clinician<br>deems appropriate | Give as soon as diagnosis of anaphylaxis is<br>suspected | 1:1000 concentration<br>0.01mg/kg OR 0.13mg<br>pediatric autoinjectable<br>(maximum 0.5mg/mg per<br>dose) |
| PATIENT<br>POSITION | | | | <ul> <li>Place patient in supine position and elevate<br/>lower extremities when there is concern for<br/>hemodynamic compromise.</li> </ul> | |
| OXYGEN | Consider 8-10 L/min<br>initially, may titrate<br>using pulse oximetry<br>as guide | Appropriate to<br>patient condition<br>– i.e. nasal canula<br>or mask | | Especially appropriate for prolonged and<br>severe reactions | Titrated using pulse oximetry as guide |
| INTRAVENOUS<br>FLUIDS | Crystalloid Solution,<br>preferably normal<br>saline (NS)<br>1 to 2 liters bolus | Intravenous | 5-10 ml/kg in the<br>first 5 minutes.<br>Colloid solution: 500<br>ml rapidly, followed<br>by slow infusion. | Caution for volume overload advised for patients with history of CHF Intraosseous access infusion can be used if IV access is unsuccessful (must use infusion pump, pressure bag, or manual pressure to overcome venous resistance) | 20-30 ml/kg in the first hour |
| INHALED<br>β2<br>ADRENERGIC<br>AGONISTS | Albuterol sulfate 2.5<br>mg/3ml unit dose or<br>Xopenex<br>(levalbuterol HCL)<br>1.25 mg/3ml unit<br>dose | Per Nebulizer via<br>mouth-piece or<br>mask as tolerated. | Delivered over 5-13<br>minutes and<br>continued as<br>necessary for<br>bronchospasm | Used when bronchospasm does not<br>respond to epinephrine | 0.15 mg/kg (minimum dose<br>2.5 mg) every 20 minutes for<br>3 doses then 0.15-0.3 mg/kg<br>(not to exceed 10 mg) every<br>1-4 hours as needed or 0.5<br>mg/kg/hour by continuous<br>nebulization |
| GLUCAGON | 1 to 5 mg IV over 5<br>minutes | Intravenous (Glucagon administered as IV push should be reconstituted with 1 ml sterile water for injection or sterile water for reconstitution) | If no response following IVP consider IV infusion, 0.05-0.1 mg/kg/h OR 1 – 5 mg/hr titrated to clinical response | Used if epinephrine is not effective in patients taking β-blockers (may reverse refractory bronchospasm and hypotension) Isotonic volume expansion may also be necessary (in some cases up to 7 L) Protection of the airway is important since glucagon can cause vomiting and risk aspiration (place in lateral recumbent position to protect airway) | 20-30 μg/kg IV x1<br>(maximum 1 mg) |
| EPINEPHRINE<br>IV | 1:100,000 solution<br>(0.1 mg [1 ml of<br>1:1000] in 100 ml<br>saline) | Intravenous | Initial rate of 30-100 ml/hr (5-15 µg/min) per infusion pump, titrate for hemodynamic response | Used in patients with poor response to IM/SQ Epinephrine Used only in profoundly hypotensive patients not responding to IV volume replacement. Every minute VS and EKG monitoring should be considered | 0.1 μg/kg/min [0.6 X body<br>weight (in kg) = # of mg<br>diluted to total 100 ml saline;<br>then 1 ml/h delivers 0.1<br>μg/kg/min] |
| VASOPRESSOR | Dopamine (400 mg in<br>300 ml of 5%<br>Dextrose) | Intravenous | 2-20 µg/kg/min,<br>titrated to maintain<br>systolic > 90 mm Hg | Used if epinephrine and volume expansion<br>fail to alleviate hypotension. Transfer to hospital ASAP | 2-20 μg/kg/min (6 X body<br>weight (in kg) = # of mg<br>diluted to total 100 ml saline;<br>then 1 ml/h delivers 1<br>μg/kg/min] |



| | | hypotension) | | | |
|---|---|---|---|---|---|
| H2<br>ANTIHISTAMINE | Famotidine (Pepcid)<br>20 mg or ranitidine<br>1mg/kg (max 50mg) | Intravenous<br>(10 mg/ml,<br>undiluted) | Administer each 20<br>mg or fraction<br>thereof over at least<br>2 minutes IV push | Side effects: headache, dizziness, constipation, diarrhea. Confusion increased in patients > 50 years old; thought to be associated with renal or hepatic impairment | 0.25 - 0.5 mg/kg (maximum<br>dose 40 mg/day) |
| CORTICO-<br>STEROID | Methylprednisolone<br>sodium succinate<br>(solumedrol)<br>IV – 40-125mg q 4-6<br>hours;<br>Status asthmaticus –<br>0.5-1mg/kg q6 hours | IV push Oral can be considered for risk of biphasic reaction, data inconclusive, doses vary | IV push doses<br>administered over 2<br>to 3 minutes | Not effective for acute treatment of<br>anaphylaxis, but may prevent protracted<br>anaphylaxis No conclusive evidence for prevention of<br>biphasic response | Children <12 years 0.5 – 1.7 mg/kg/day divided q6 – 12h. Status asthmaticus – 0.5- 1mg/kg q6 hours |

## 7. <u>Study Intervention Discontinuation and Participant Discontinuation/Withdrawal</u>

### 7.1 Discontinuation of Study Intervention

Criteria for discontinuing oral immunotherapy in a subject will include:

- Subject nonadherence to OIT, specifically defined by 12 (approximately 10%) nonconsecutive missed doses.
- A life-threatening adverse reaction to OIT, specifically a grade 4 reaction as defined by the Consortium of Food Allergy Research (CoFAR) criteria. See table in Section 8.3.3.1.
- Symptoms suggestive of Eosinophilic Esophagitis of (EoE) i.e. difficulty swallowing, chest pain, persistent heart burn, upper abdominal pain, and/or no response to gastroesophageal reflux disease (GERD) medication

Symptoms suggestive of Eosinophilic Esophagitis (EoE) will prompt discontinuation of oral immunotherapy and begin once weekly symptom monitoring phone calls with study staff. If symptoms fail to resolve after 1 month off therapy, consultation with Gastroenterology will be considered for further evaluation and management.

Discontinuation from oral immunotherapy does not mean discontinuation from the study, and remaining study procedures should be completed as indicated by the study protocol. If a clinically significant finding is identified (including, but not limited to changes from baseline) after enrollment, the investigator or qualified designee will determine if any change in participant management is needed. Any new clinically relevant finding will be reported as an adverse event (AE).

The data to be collected at the time of study intervention discontinuation will include the following:

- Skin prick test to peanut
- Peanut slgE, peanut component panel, and peanut lgG4

### 7.2 Participant Discontinuation/Withdrawal from the Study

Participants are free to withdraw from participation in the study at any time upon request. Subjects may withdraw from the study for the following anticipated reasons

- Adverse events related to OIT
  - Chronic or recurrent GI symptoms
  - Acute hypersensitivity reactions
  - Chronic or recurrent cutaneous symptoms
- Social reasons: time constraints, transport
- Principal Investigator temporarily suspends or prematurely discontinues study participation. The
  date and reason for discontinuation must be documented (e.g. non-compliance). Every effort
  should be made to complete the appropriate assessments.
- Pregnancy during the course of the study for a child-bearing participant
- The investigator considers it, for safety reasons, to be in the best interest of the subject.
- Disease progression
  - o Worsening asthma that requires increasing therapy such that exclusion criteria are met

The reason for subject discontinuation or withdrawal from the study will be recorded on the Case Report Form (CRF). Subjects who sign the informed consent form and are enrolled but do not receive the study intervention may be replaced. Subjects who sign the informed consent form, and are enrolled and receive the study intervention, and subsequently withdraw, or are withdrawn or discontinued from the study, will not be replaced.

### 7.3 Lost to Follow-up

A participant will be considered lost to follow-up if he or she fails to return for 2 scheduled visits and is unable to be contacted by the study site staff.

The following actions must be taken if a participant fails to return to the clinic for a required study visit:

- The site will attempt to contact the participant and reschedule the missed visit within 1 week for an updosing visit or within 1 month for a follow up visit and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain if the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee will make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record or study file.
- Should the participant continue to be unreachable, he or she will be considered to have withdrawn from the study with a primary reason of lost to follow-up.

### 8. Study Assessments and Procedures

### **8.1 Efficacy Assessments**

**Procedures** 

Skin tests: Skin testing to peanut will be performed at the visits specified in the SoA (section 1.3). Skin testing will include skin prick with peanut exact (1:20 w/v, Greer), negative control (saline) and positive control (histamine).

Laboratory tests: Blood samples will be collected at the visits specified in the SoA. Blood work will include peanut specific IgE concentration, peanut component testing (peanut specific IgE concentration for Ara h 1, 2, 3, 8 and 9), and peanut specific IgG4 concentration. The peanut sIgE and peanut component panel will be sent to the Cleveland Clinic main laboratory. The peanut specific IgG4 will be sent to Mayo Clinic laboratories. The laboratories used will supply a list of reference ranges and units of the laboratory parameters.

Volume of blood to be collected:

Peanut specific IgE concentration 0.5 mL
Peanut component panel 0.6 mL
Peanut IgG4 concentration 0.5 mL
Total 1.6 mL

### **8.2 Safety and Other Assessments**

Screening to ensure all subjects meet the inclusion criteria and do not meet any exclusion criteria will be performed within 1 month of the initial oral food challenge visit. At Visit 1, the physician and participant will review and update the patient's Food Allergy & Anaphylaxis Emergency Care Plan. This plan will outline the recommended treatment in case of an allergic reaction occurs during their enrollment in the study. This plan is signed by a physician, and includes emergency contact information. In addition, each study visit will include obtaining a brief interim history to ensure that no potential augmenting factors, such as viral illness, are present at the time of study drug or control drug administration. Vital signs, a targeted physical exam and conmed review will be performed prior to any study drug administration for the same purposes.

Study visit evaluation:

Brief interim history

Discussion of any interim AEs

Vital signs: Temperature, Heart Rate, Respiratory Rate

Physical Exam: Targeted assessment of General Appearance, HEENT, Cardiac, Respiratory, Abdominal,

and Skin

### 8.3 Adverse Events and Serious Adverse Events

### 8.3.1 Definition of Adverse Event

Adverse event means any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related (21 CFR 312.32 (a)).

The CoFAR (the consortium of Food Allergy research) scale will be referenced to assess SAEs/AEs related or possibly related to an allergic reaction. CTCAE (Common Terminology Criteria for Adverse Events) version 5.0 will be referenced for SAEs/AEs that are not related to allergic reactions and are therefore not listed in the CoFAR scale.

### 8.3.2 Definition of Serious Adverse Events (SAE)

An adverse event (AE) or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home or hypotension not responsive to treatment with epinephrine.

### 8.3.3 Classification of an Adverse Event

### 8.3.3.1 Severity of an Event

All adverse events will be graded in severity utilizing criteria specifically developed by the Consortium of Food Allergy Research.<sup>27</sup> These criteria are widely accepted and applied to OIT clinical trials.

| Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|
| Mild | Moderate | Severe | Life threatening | Death |
| Transient or mild | Symptoms that produce | Marked limitation in | Extreme limitation in | Death |
| discomforts (< 48 | mild-to-moderate | activity, some | activity, significant | |
| hours), no or minimal | limitation in activity, | assistance usually | assistance required; | |
| medical | some assistance may be | required; medical | significant | |
| intervention/therapy | needed; no or minimal | intervention/therapy | medical/therapy. | |
| required. These | intervention/therapy is | required, | Intervention is | |
| symptoms may | required. | hospitalization is | required; | |
| include | Hospitalization is | possible. Symptoms | hospitalization is | |
| pruritus, swelling or | possible. These | may include | probable. Symptoms | |
| rash, abdominal | symptoms may include | bronchospasm with | may include persistent | |
| discomfort or other | persistent hives, | dyspnea, severe | hypotension and/or | |
| transient symptoms. | wheezing without | abdominal pain, throat | hypoxia with resultant | |
| | dyspnea, abdominal | tightness with | decreased level of | |
| | discomfort/increased | hoarseness, and | consciousness | |
| | vomiting or other | transient hypotension | associated with | |
| | symptoms. | among others. | collapse and/or | |
| | | Parenteral | incontinence or other | |
| | | medication(s) are | life-threatening | |
| | | usually indicated. | symptoms | |

### 8.3.3.2 Relationship to Study Intervention

All adverse events (AEs) must have their relationship to study intervention assessed by the clinician who examines and evaluates the participant based on temporal relationship and his/her clinical judgment.

The degree of certainty about causality will be graded using the categories below. In a clinical trial, the study product must always be suspect.

- Definitely Related There is clear evidence to suggest a causal relationship, and other possible
  contributing factors can be ruled out. The clinical event, including an abnormal laboratory test
  result, occurs in a plausible time relationship to study intervention administration and cannot be
  explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the
  study intervention (dechallenge) should be clinically plausible. The event must be
  pharmacologically or phenomenologically definitive, with use of a satisfactory rechallenge
  procedure if necessary.
- Probably Related There is evidence to suggest a causal relationship, and the influence of other
  factors is unlikely. The clinical event, including an abnormal laboratory test result, occurs within
  a reasonable time after administration of the study intervention, is unlikely to be attributed to
  concurrent disease or other drugs or chemicals, and follows a clinically reasonable response on
  withdrawal (dechallenge). Rechallenge information is not required to fulfill this definition.
- Potentially Related There is some evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of the trial medication). However, other factors may have contributed to the event (e.g., the participant's clinical condition, other concomitant events). Although an AE may rate only as "possibly related" soon after discovery, it can be flagged as requiring more information and later be upgraded to "probably related" or "definitely related", as appropriate.
- Unlikely to be related A clinical event, including an abnormal laboratory test result, whose temporal relationship to study intervention administration makes a causal relationship improbable (e.g., the event did not occur within a reasonable time after administration of the study intervention) and in which other drugs or chemicals or underlying disease provides plausible explanations (e.g., the participant's clinical condition, other concomitant treatments).
- Not Related The AE is completely independent of study intervention administration, and/or
  evidence exists that the event is definitely related to another etiology. There must be an
  alternative, definitive etiology documented by the clinician

### 8.3.3.3 Expectedness

An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the risk information previously described for the study intervention.

### 8.3.4 Time Period and Frequency for Event Assessment and Follow-up

The occurrence of an adverse event (AE) or serious adverse event (SAE) may come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care, or upon review by a study monitor.

All AEs including local and systemic reactions not meeting the criteria for SAEs will be captured on the appropriate case report form (CRF). Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product (assessed only by those with the training and authority to make a diagnosis), and time of resolution/stabilization of the event. All AEs occurring while on study must be documented appropriately regardless of relationship. All AEs will be followed to adequate resolution.

Any medical condition that is present at the time that the participant is screened will be considered as baseline and not reported as an AE. However, if the study participant's condition deteriorates at any time during the study, it will be recorded as an AE.

Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode.

All reportable events will be recorded with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization.

### 8.3.5 Adverse Event Reporting

An independent Data Safety Monitoring Board (DSMB) will be utilized during the study. The DSMB will consist of 2 Board Certified Allergy/Immunology physicians who are not participating in the study and do not have any conflicts of interest as well as 1 pediatric physician of another specialty. The DSMB will meet prior to initiation of the study, following the enrollment of the 6<sup>th</sup> subject, and then quarterly during the course of the study.

### 8.3.6 Serious Adverse Event Reporting

The study clinician will immediately report to the sponsor any serious adverse event, whether or not considered study intervention related, including those listed in the protocol or investigator brochure and must include an assessment of whether there is a reasonable possibility that the study intervention caused the event. Study endpoints that are serious adverse events (e.g., all-cause mortality) must be reported in accordance with the protocol unless there is evidence suggesting a causal relationship between the study intervention and the event (e.g., death from anaphylaxis). In that case, the investigator must immediately report the event to the sponsor.

All serious adverse events (SAEs) will be followed until satisfactory resolution or until the site investigator deems the event to be chronic or the participant is stable. Other supporting documentation of the event may be requested by the study sponsor and should be provided as soon as possible.

The study sponsor is responsible for notifying the Food and Drug Administration (FDA) of any unexpected fatal or life-threatening suspected adverse reaction as soon as possible, but in no case later than 7 calendar days after the sponsor's initial receipt of the information. In addition, the sponsor must notify FDA and all participating investigators in an Investigational New Drug (IND) safety report of potential serious risks, from clinical trials or any other source, as soon as possible, but in no case later than 15 calendar days after the sponsor determines that the information qualifies for reporting

### 8.3.7 Reporting Events to Participants

All anticipated AEs will involve overt symptoms and thus be readily apparent to the subjects and their families. When an AE occurs during a study visit, the nature and severity of the AE as well as the implications for ongoing treatment will be discussed by a physician investigator with the subject and parents/guardians. This discussion will take place after any potential treatment is administered and the subject is deemed medically stable but prior to end of the study visit.
When an AE occurs at home, the nature and severity of the AE as well as the implications for ongoing treatment will be discussed by a physician investigator with the subject and parents/guardians via phone. If a study visit is deemed appropriate to further manage the AE or for further discussion of the AE, then additional discussion will take place at this time.

#### 8.3.8 Events of Special Interest

This is not applicable to our study.

#### 8.3.9 Reporting of Pregnancy

If a pregnancy were to occur during the course of the study, the subject would be withdrawn from the study. The pregnancy would be reported the PRRC and IRB at the Cleveland Clinic. The subject would be referred to an appropriate physician (OB/Gyn) for further management.

#### 8.4 Unanticipated Problems

### 8.4.1 Definition of Unanticipated Problems (UP)

The Office for Human Research Protections (OHRP) considers unanticipated problems involving risks to participants or others to include, in general, any incident, experience, or outcome that meets all of the following criteria:

- Unexpected in terms of nature, severity, or frequency given (a) the research procedures that are
  described in the protocol-related documents, such as the Institutional Review Board (IRB)approved research protocol and informed consent document; and (b) the characteristics of the
  participant population being studied;
- Related or possibly related to participation in the research ("possibly related" means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and
- Suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

#### 8.4.2 Unanticipated Problem Reporting

The investigator will report unanticipated problems (UPs) to the reviewing Institutional Review Board (IRB) and to the lead principal investigator (PI). The UP report will include the following information:

- Protocol identifying information: protocol title and number, PI's name, and the IRB project number;
- A detailed description of the event, incident, experience, or outcome;
- An explanation of the basis for determining that the event, incident, experience, or outcome represents an UP;
- A description of any changes to the protocol or other corrective actions that have been taken or are proposed in response to the UP.

To satisfy the requirement for prompt reporting, UPs will be reported using the following timeline:

• UPs that have serious impact or require a change to the protocol will be reported to the IRB and to the study sponsor within 10 days of the investigator becoming aware of the event.

All UPs should be reported to appropriate institutional officials (as required by an institution's
written reporting procedures), the supporting agency head (or designee), and the Office for
Human Research Protections (OHRP). The reporting timeline for UPs that do not have serious
impact or require a change to the protocol will be the time of continuing renewal with the IRB.

#### 8.4.3 Reporting Unanticipated Problems to Participants

Should unanticipated problems arise that have serious impact to the protocol or to the safety of participants, participants will be notified based on the opinion of the IRB once the UP has been reviewed.

### 9. Statistical Considerations

#### 9.1 Statistical Hypothesis

We will obtain observation data on patients receiving boiled peanut oral immunotherapy which has not yet been well described in human trials. We will compare with proportion of patients successfully desensitized as defined by meeting the primary endpoint with the expected placebo rate. The null hypothesis is that the proportion of patients successfully desensitized by boiled peanut oral immunotherapy will not be greater than the expected 20% that has been previously published as the proportion of patients successfully meeting the primary endpoint in OIT studies (which aligns with the expected 20% that would naturally "outgrow" a peanut allergy). If we reject this null hypothesis, we will be able to conclude that the proportion of successfully desensitized by boiled peanut therapy is greater than placebo. For the safety aspect of the study we will be comparing the historical SAEs/AEs of patients who received OIT with roasted peanuts and compare them with the patients enrolled in this study for the rate of occurrence and severity of the SAEs/AEs observed.

#### 9.2 Sample Size Determination

The sample of 10 patients will provide >90% power to determine the expected success rate (80%) is greater than a theoretical placebo rate (20%).

### 9.3 Populations for Analysis

Both an Intentional-to-Treat (ITT) and per-protocol analysis will be performed.

#### 9.4 Statistical Analysis

Descriptive statistics will be used to summarize the data. Categorical variables will be presented as number and percentage of total patients. Continuous variables will be summarized using mean, standard deviation, median and [Q1, Q3]. The proportion of patients with successful consumption of peanut protein without symptoms (primary endpoint), will be tested to determine whether the proportion differs from 0.2 (20%) (the expected success rate in a theoretical placebo group).

## **10.Supporting Documentation and Operational Considerations**

#### 10.1 Regulatory, Ethical and Study Oversight Considerations

10.1.1 Informed Consent Process

10.1.1.1 Consent/Assent and Other Informational Documents Provided to Participants
Consent forms describing in detail the study intervention, study procedures, and risks are given to the participant and written documentation of informed consent is required prior to starting intervention/administering study intervention. The following consent materials are submitted with this protocol:

- Informed Consent
- Informed Assent

#### 10.1.1.2 Consent Procedures and Documentation

Informed consent is a process that is initiated prior to the individual and parent/guardian's agreeing to participate in the study and continues throughout the individual's study participation. Consent forms will be Pediatric ResearchReview Committee (PRRC) and Institutional Review Board (IRB)-approved and the participant and/or parent/guardian will be asked to read and review the document. The investigator will explain the research study to the participant and parent/guardian and answer any questions that may arise. A verbal explanation will be provided in terms suited to the participant and parent/guardian's comprehension of the purposes, procedures, and potential risks of the study and of their rights as research participants. Participants and parents/guardians will have the opportunity to carefully review the written consent form and ask questions prior to signing. The participants and parents/guardians should have the opportunity to discuss the study with their family or surrogates or think about it prior to agreeing to participate. The participant's parent/guardian will sign the informed consent document prior to any procedures being done specifically for the study. Participants and parents/guardians must be informed that participation is voluntary and that they may withdraw from the study at any time, without prejudice. A copy of the informed consent document will be given to the participant's parent/guardian for their records. The informed consent process will be conducted and documented in the source document (including the date), and the form signed, before the participant undergoes any study-specific procedures. The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study

#### 10.1.2 Study Discontinuation and Closure

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to <study participants, investigator, funding agency, the Investigational New Drug (IND) or Investigational Device Exemption (IDE) sponsor and regulatory authorities>. If the study is prematurely terminated or suspended, the Principal Investigator (PI) will promptly inform study participants, the Institutional Review Board (IRB), and sponsor and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Demonstration of efficacy that would warrant stopping
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Determination that the primary endpoint has been met
- Determination of futility

Study may resume once concerns about safety, protocol compliance, and data quality are addressed, and satisfy the sponsor, IRB and/or Food and Drug Administration (FDA).

#### 10.1.3 Confidentiality and Privacy

Participant confidentiality and privacy is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their interventions. This confidentiality is extended to cover testing of biological samples and genetic tests in addition to the clinical information relating to participants. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

All research activities will be conducted in as private a setting as possible.

The study monitor, other authorized representatives of the sponsor, representatives of the Institutional Review Board (IRB), regulatory agencies or pharmaceutical company supplying study product may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

The study participant's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB, Institutional policies, or sponsor requirements.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at within RedCap Cloud. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by clinical sites and by CRU research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived within RedCap Cloud.

### 10.1.4 Future Use of Stored Specimens and Data

Data will be maintained on RedCap Cloud per institute policy. Stored specimens will be discarded after analysis per Cleveland Clinic Laboratory policy.

10.1.5 Key Roles and Study Governance Principal Investigator Jaclyn Bjelac, MD Staff, Pediatric Allergy and Immunology Cleveland Clinic 9500 Euclid Ave/A120 Cleveland, OH 44195

Medical Monitor Clinical Research Unit

## 11. References

- 1. Bunyavanich et al. Letter to the Editor: Peanut allergy prevalence among school age children in a US cohort not selected for any disease. J Allergy Clin Immunol. 2014 Sep;134(3):753-5.
- 2. Bock SA, Muñoz-Furlong A, Sampson HA. Fatalities due to anaphylactic reactions to foods. J Allergy Clin Immunol. 2001 Jan;107(1):191-3.
- 3. Sicherer, SH and Sampson, HA. Food allergy: A review and update on epidemiology, pathogenesis, diagnosis, prevention, and management. J Allergy Clin Immunol. 2018 Jan;141(1):41-58.
- 4. Primeau MN, Kagan R, Joseph L, et al. The psychological burden of peanut allergy as perceived by adults. Clin Exp Allergy. 2000 Aug;30(8):1135-43.
- 5. Sicherer SH, Noone SA, Muñoz-Furlong A. The impact of childhood food allergy on quality of life. Ann Allergy Asthma Immunol. 2001 Dec;87(6):461-4.
- 6. Sampson HA et al. Food allergy: A practice parameter update-2014. J Allergy Clin Immunol. 2014 Nov;134(5):1016-25.
- 7. Wood, RA. Food allergen immunotherapy: current status and prospects for the future J Allergy Clin Immunol. 2016 Apr;137(4):973-982.
- 8. Jones, SM, et al. Clinical efficacy and immune regulation with peanut oral immunotherapy. J Allergy Clin Immunol. 2009 Aug;124(2):292-300.
- 9. Blumenchen, K et al. Oral peanut immunotherapy in children with peanut anaphylaxis. J Allergy Clin Immunol. 2010 Jul;126(1):83-91.
- 10. Hofmann, AM, et al. Safety of a peanut oral immunotherapy protocol in children with peanut allergy. J Allergy Clin Immunol. 2009 Aug;124(2):286-91.
- 11. Varshney, P, et al. A randomized controlled study of peanut oral immunotherapy: clinical desensitization and modulation of the allergic response. J Allergy Clin Immunol. 2011 Mar;127(3):654-60.
- 12. Anagnostou K, et al. Efficacy and safety of high-dose peanut oral immunotherapy with factors predicting outcome. Clin Exp Allergy. 2011 Sep;41(9):1273-81.
- 13. Anagnostou K, et al. Assessing the efficacy of oral immunotherapy for the desensitisation of peanut allergy in children (STOP II): a phase 2 randomised controlled trial. Lancet. 2014 Apr 12;383(9925):1297-304.
- 14. Vickery, VP, et al. Sustained unresponsiveness to peanut in subjects who have completed peanut oral immunotherapy. J Allergy Clin Immunol. 2014 Feb;133(2):468-75.
- 15. Narisety, SD, et al. A randomized, double-blind, placebo-controlled pilot study of sublingual versus oral immunotherapy for the treatment of peanut allergy. J Allergy Clin Immunol. 2015 May;135(5):1275-82.
- 16. Vickery, VP, et al. Early oral immunotherapy in peanut-allergic preschool children is safe and highly effective. J Allergy Clin Immunol. 2017 Jan;139(1):173-181.
- 17. Maleki SJ, Chung SY, Champagne ET, Raufman JP. The effects of roasting on the allergenic properties of peanut proteins. J Allergy Clin Immunol. 2000 Oct;106(4):763-8.
- 18. Beyer K, Morrow E, Li XM, et al. Effects of cooking methods on peanut allergenicity. J Allergy Clin Immunol. 2001 Jun;107(6):1077-81.
- 19. Tao B et al. Extended boiling of peanut progressively reduces IgE allergenicity while retaining T cell reactivity. Clin Exp Allergy. 2016 Jul;46(7):1004-14.
- 20. Turner PJ, Mehr S, et al. Letter to the Editor: Loss of allergenic proteins during boiling explains tolerance to boiled peanut in peanut allergy. J Allergy Clin Immunol. 2014; 134:751-3.

- 21. Bird, JA, et al. Efficacy and Safety of AR101 in Oral Immunotherapy for Peanut Allergy: Results of ARC001, a Randomized, Double-Blind, Placebo-Controlled Phase 2 Clinical Trial. J Allergy Clin Immunol Pract. 2018 Mar Apr;6(2):476-485.
- 22. United States Department of Agriculture. USDA National Nutrient Database for Standard Reference, release 21. 2002. Available at: http://ars.usda.gov/Services/docs.htm?docid=17477.
- 23. Virkud YV, et al. Novel baseline predictors of adverse events during oral immunotherapy in children with peanut allergy. J Allergy Clin Immunol. 2017 Mar;139(3):882-888
- 24. Klemans RJ, et al. Ara h 2 is the best predictor for peanut allergy in adults. J Allergy Clin Immunol Pract. 2013 Nov-Dec;1(6):632-8.
- 25. Wasserman, RL, et al. Oral Immunotherapy for Peanut Allergy: Multipractice Experience With Epinephrine-treated Reactions. J Allergy Clin Immunol Pract. 2014 Jan-Feb;2(1):91-6.
- 26. Rigbi, NE, et al. Changes in patient quality of life during oral immunotherapy for food allergy. Allergy. 2017 Dec;72(12):1883-1890.
- 27. Factor JM et al. Effect of oral immunotherapy to peanut on food-specific quality of life . Ann Allergy Asthma Immunol 109 (2012) 348-352.
- 28. Burks, AW et al. Oral immunotherapy for treatment of egg allergy in children N Engl J Med. 2012 Jul 19;367(3):233-43.

# 12. Supplements

## 12.1 Food Allergy Quality of Life Questionnaire for Parents (1-12 years old)

Supplement 1 A

#### Food Allergy Quality of Life Questionnaire for Parents (children 1-12 years old)

Instructions: The questions below are about the influence of food allergy on your child's quality of life. If is important that all questions be completed.

Answer every question by putting an 'v' in the proper box. You may choose from the following answers:

| Answer every question by putting an 'x' in the proper box. You may choose from the folio | | | | | | | _ |
|---|---|---|---|---|---|---|---|
| | 1<br>Not | 2<br>Barely | 3<br>A little | 4<br>Fairly | 5<br>Quite | 6<br>Very | 7<br>Extremel |
| Because of food allergy, my child feels | | , | | , | - | , | |
| 1. Different from other children | | | | | | | |
| Because of food allergy, my child has been negatively affected by | | | | | | | |
| <ol><li>Receiving more attention than other children of his/her age</li></ol> | | | | | | | |
| <ol><li>Having to grow up more quickly than other children of his/her age</li></ol> | | | | | | | |
| 4. His/her environment being more restricted than other children of his/her age | | | | | | | |
| Because of food allergy, my child | | | | | | | |
| 5. Experiences physical distress | | | | | | | |
| 6. Experiences emotional distress | | | | | | | |
| 7. Is more anxious in general than other children of his/her age | | | | | | | |
| 8. Is more cautious in general than other children of his/her age | | | | | | | |
| 9. Is not as confident as other children of his/her age in social situations | | | | | | | |
| 10. Wishes his/her food allergy would go away | | | | | | | |
| 11. Has a lack of variety in his/her diet | | | | | | | |
| Because of food allergy, my child feels | | | | | | | |
| 13. Anxious about food | | | | | | | |
| 13. Afraid to try unfamiliar foods | | | | | | | |
| 14. Concerned that I am worried that he/she will have a reaction to food | | | | | | | |
| 15. Frustrated by dietary restrictions | | | | | | | |
| 16. Left out of activities involving food | | | | | | | |
| Because of food allergy, my child's ability to take part has been limited | | | | | | | |
| 17. By anxiety when going to new places | | | | | | | |
| 18. By concern that he/she must always be cautious about food | | | | | | | |
| 19. By anxiety when eating with unfamiliar adults/children | | | | | | | |
| 20. In social activities in other people's houses (sleepovers, parties, playtime) | | | | | | H | |
| 21. In preschool/school events involving food (class parties/treats/lunchtime) 22. Being upset that family social outings have been limited by food allergy | | 님 | | | | 님 | |
| , , , | | | | | | H | |
| 23. By frustration from social restrictions<br>24. Restaurants we can safely go to as a family | | | | | | 님 | |
| | ΙH | | | | H | H | H |
| 25. Holiday destinations we can safely go to as a family | " | | | | | | |
| How troublesome did you find side effects of oral immunotherapy (OIT)? | | | | | | | |

## 12.2 Food Allergy Quality of Life Questionnaire for Parents (13-16 years old)

Supplement 1B

#### Food Allergy Quality of Life Questionnaire for Adolescents (13-16 years old)

Instructions: The questions below are about the influence of food allergy on your quality of life. If is important that all questions be completed. Answer every question by putting an 'x' in the proper box. You may choose from the following answers:

| | 1<br>Not | 2<br>Barely | 3<br>A little | 4<br>Fairly | 5<br>Quite | 6<br>Very | 7<br>Extremely |
|---|---|---|---|---|---|---|---|
| How troublesome do you find it, because of your food allergy, that you 1. Must always be alert as to what you are eating? 2. Are able to eat fewer products 3. Are limited by the products you can buy 4. Must read labels 5. Are less easily able to spontaneously accept an invitation to stay for a meal? 6. Are les able to taste or try various products when eating out? 7. Must check yourself whether you can eat something when eating out? 8. Hesitate eating a product when you have doubts about it? 9. Must refuse treats at school or work? 10. That you have to explain to people around you that you have a food allergy? 11. Have the feeling that you have less control of what you eat when eating out? 12. Must carry an epinephrine auto injector? 13. Must be careful about touching certain foods 14. That the ingredients of a product change? 15. That the label states, "may contain traces of peanut?" 16. That the labeling of the bulk packaging (for example box or bag) is different than the individual packages? | | | 000000000000000000000000000000000000000 | | | | |
| 17. That during social activities others can eat the food to which you are allergic? 18. That during social activities your food allergy is not taken into account enough? | | | | | | | |
| How <i>frightened</i> are you, because of your food allergy 19. Of an allergic reaction? 20. Of unintentionally eating the wrong food? 21. To eat something you have never before? | | | | | | | |
| Please answer the following questions: 22. How <i>discouraged</i> do you feel during an allergic reaction? | | | | | | | |
| After completion of study only: 23. How troublesome did you find side effects of oral immunotherapy (OIT)? | | | | | | | |

# 12.3 Dosing/Adverse Events Recording Sheet

Supplement 2

## **Dosing/Adverse Events Recording Sheet**

Patient Name Number:

| Date | Dose | - | Time of Dose | | | |
|---|---|---|---|---|---|---|
| Any Reaction? | □ Yes | □ No | | | | |
| If yes | | | | | | |
| Symptoms of Reaction? (checkall that apply) | ☐ Rash/hives | ☐ Lip/Mouth<br>Itching | ☐ Nausea/Upset<br>Stomach | ☐ Vomiting | ☐ Cough/<br>Wheeze | ☐ Other: Please comment |
| Treatment Required? | □ No | ☐ Yes | If yes, what? | ☐ Antihistamines | ☐ Albuterol | ☐ Epinephrine |
| How soon after dose did symptoms begin? | ☐ Within 5-10 minutes | ☐ 10-60 minutes | ☐ 60-120<br>minutes | □ >120 minutes | | |
| Location of rash, if present (check all that apply) | ☐ Face | ☐ Neck/Chest | ☐ Arms and/or legs | ☐ Stomach and/or back | | |
| How long were symptoms present before treatment was given? | ☐ < 10 minutes | ☐ 10-30 minutes | ☐ 30-60 minutes | □ > 60 minutes | | |
| How many doses of treatment were given? | □ 1 | □ 2 | ☐ 3 or more | | | |
| How long did symptoms last? | □ <10 minutes | ☐ 10-60 minutes | ☐ 60-120<br>minutes | □ >120 minutes | | |
| Any other comments? | | · | | | | |

### **SUMMARY OF CHANGES**

Please provide a list of changes from the previous approved version of the protocol starting at IRB approval. This table will remain blank until initial IRB approval. The list shall be a brief overview. When appropriate, a brief justification for the change should be included. This is a running list for the life of the study.

| Protocol<br>Date | Section | Change |
|---|---|---|
| 04.02.2019 | Footer and PSP | Changed Version number and version date to 4.0 and 4-2-19 respectively |
| | 6. Study Intervention | All references to "UH Lerner Tower Kitchen" were replaced with "UH Dahms Clinical Research Unit" |
| | 6. Study Intervention | The onging post study OIT maintenance period was changed to being optional for study participants and is not paid for by the study. |
| | 8.2 Study Assessments and Procedures | At Visit 1, the physician and participant will review and update the patient's Food Allergy & Anaphylaxis Emergency Care Plan. Conmed review also added before each dose escalation |
| | PSP and section 8.3.9 | Changed PIRC (Pediatric Institute Review Committee) to PRRC (Pediatric Research Review Committee) |
| | Inclusion criteria | Added the additional language "within a 12 month period of study enrollment" in the inclusion criteria requiring Evidence of IgE mediated peanut hypersensitivity |
| | 1.3 Schedule of activities and section 6.1 | Added Urine Pregnancy |
| | 6.2 IP dispensing | Remove randomize to treat and place a blinded label on jar from. |
| | Section 7.2 | Added additional reasons for discontinuation |
| | 1.3 Schedule of activities | Changed Adverse event review to AE review, added Study drug compliance and conmed assessment lines |

| Protocol<br>Date | Section | Change |
|---|---|---|
| | 8.3.1 | The CoFAR and CTCAE are mentioned as the scales that will be used to assess SAEs/AEs |
| | 8.4.2 and 8.4.3 | Rewording of reporting requirements and timelines |
| 05.28.2019 | PSP and footer | Updated amendment # and version date |
| | Schedule of events, table #4 and table #5 | Added spirometry and peak flow measure to study visits |
| | 9.1 Statistical Hypothesis | Added language in regards to safety hypothesis |
| 10.01.2019 | PSP and footer | Updated amendment # and version date |
| | Schedule of Events section 1.3 and section 6.1 | Added additional urine pregnancy at visit 10 |
| | Schedule of Events section 1.3 | Added language on spirometry being done at investigators discretion at enrollment as well visit 10 |
| | Section 6.1 | Clarified that the location of the skin prick test must be the same throughout the study |
| | Section 6.1 and table 7 | Added a 25 mg dose in DBOFC as well as clarification that additional smaller doses may be necessary on a patient by patient basis depending on the results of the initial OFC |
| | Section 6.1 | In build-up phase a dose double the size of the highest tolerated dose in the initial escalation may be used before the patient can be entered into the build-up phase schedule |
| 02.12.2020 | Footer | Updated protocol version date and amendment number |
| | PSP | Added signature line for sponsor |
| | Inclusion criteria | Added verbiage to inclusion criteria #2 "or a high level of suspicion based on testing at the discretion of the investigator." |

| Protocol<br>Date | Section | Change |
|---|---|---|
| | Initial dose escalation (Table 5) | Removed the first 2 doses in the initial dose escalation (0.1 and 0.2 milligrams of peanut protein). Added a 4mg dose to be given at +90 minutes. Adjusted time for 6mg dose to +120 minutes |